CLINICAL TRIAL: NCT06928857
Title: Pilot Study on the Effects Induced by an Electromyographic-controlled Functional Electrical Stimulator (FitFES) for Upper Limb Rehabilitation in Post-stroke Patients
Brief Title: Study on the Effects of an EMG-controlled Functional Electrical Stimulator for Upper Limb for Post-stroke Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: Istituto Italiano di Tecnologia (Other); Ospedale Policlinico San Martino (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RAISE-FITFES-RCT
Record Dates: First submitted 2025-01-29; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Stroke
Keywords: EMG-controlled Functional Electrical Stimulation; Stroke rehabilitation; Medical device
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FES group (Experimental): Subjects will use the device as need-based support to perform task-oriented exercises
  Interventions: Device: EMG-based FES rehabilitation
- CON group (Active Comparator): Subjects will perform task-oriented exercises without the support of the device
  Interventions: Other: Traditional rehabilitation

INTERVENTIONS:
Device: EMG-based FES rehabilitation — Each subject will receive 15 individual rehabilitation sessions, each lasting 60 minutes, conducted 3 to 5 times per week over a period of 5 to 3 weeks, depending on the weekly frequency. Each participant will perform task-oriented exercises while using the FitFES device.
  Arms: FES group
Other: Traditional rehabilitation — Each subject will receive 15 individual rehabilitation sessions, each lasting 60 minutes, conducted 3 to 5 times per week over a period of 5 to 3 weeks, depending on the weekly frequency. Each participant will perform task-oriented exercises.
  Arms: CON group

SUMMARY:
Upper limb disabilities are among the most debilitating issues after a cerebral stroke. One promising approach in motor rehabilitation is the use of functional electrical stimulation (FES). This technique can be integrated into daily therapy to follow an adaptive approach, exploiting the residual capacities of patients. FES can help to stimulate the affected muscles, improve coordination and strengthen the weakened muscles, thus supporting the rehabilitation process.

DETAILED DESCRIPTION:
FitFES is a wearable and non-invasive device that provides continuous stimulation set according to the residual myoelectric activity of hemiparetic muscles. Its bioinspired functioning has been implemented to restore the neurophysiological feedback from the muscles to the central nervous system while performing voluntary movements. This study aims to assess the effects of FitFES device on upper limb motor rehabilitation of post-stroke subjects, compared to traditional rehabilitation treatment. 50 post-stroke subjects will be recruited and randomized into an experimental group and a control group.

All participants will follow a 15-session rehabilitation program, and in each session they will execute task-oriented exercises. The experimental group will be assisted by the FitFES device, while the control group will perform the tasks without the device support.

Each subject will be assessed before and at the end of the rehabilitation protocol. Collected data from both groups will then be compared.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Diagnosis of first ischemic or hemorrhagic unilateral stroke for at least two weeks
* Medical Research Council score for at least one upper limb muscle greater than 0 and less than 5 (excluding extremes).
* Signed informed consent

Exclusion Criteria:

* Score at the Mini Mental State Examination (adjusted for age and schooling) < 24
* Clinical evidence in the case of visual disturbance, ideomotor apraxia, behavioral disorders, neglect, sensory, visual and auditory disturbances of severe degree or otherwise that prevent use of the device
* Major head trauma
* Cardio-respiratory or internal clinical instability
* State of pregnancy or lactation
* Severe spasticity (Ashworth > 3)
* Skin integrity problems at the interface surface with the device
* Implanted electronic devices
* Epilepsy not medically controlled
* Severe peripheral neuropathy
* Recent interventions
* Thrombosis, thrombophlebitis
* Active stent carrier less than six months
* Severe forms of arteriosclerosis, arterial circulatory disorders
* Hypertension not treated
* Cardiac arrhythmias
* Hemorrhagic disorders (hemophilia)
* Severe forms of diabetes mellitus
* Known allergy to materials making up the device or its applied parts
* Cancer or tumour disease
* Acute arthritis
* Other neurological diseases other than stroke
* Progressive muscular dystrophy
* Abdominal or inguinal hernias
* Undiagnosed back pain
* Diseases of internal organs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Action Research Arm Test (ARAT) | Baseline (T0), after 15 rehabilitation sessions (each session is 60 minutes) from 3 to 5 weeks after T0 (T1), 1-month follow-up (T2)
  The ARAT test assesses upper limb functioning through the execution of 19 tasks, divided in 4 sub-tests (grasp, grip, pinch, and gross arm movement). Each movement is scored on a 4-point ordinal scale (0=no movement, 1=movement partially performed, 2=movement completed but takes abnormally long; 3=movement performed normally). Total possible score is 57 points, with higher scores associated to best motor functioning.
Fugl-Meyer Upper Extremity scale (FM-UE) | Baseline (T0), after 15 rehabilitation sessions (each session is 60 minutes) from 3 to 5 weeks after T0 (T1), 1-month follow-up (T2)
  The Fugl-Meyer Assessment of Motor Recovery after Stroke is one of the most widely used measures of motor impairment in post-stroke hemiplegic patients, covering 5 domains (Motor fu ENnction, sensory function, balance, joint range of motion, joint pain). The assessment of upper extremity motion is performed using the Upper Extremity assessment (FM-UE), including items scored on a 3-point ordinal scale (0: cannot perform, 1: performs partially; 2: performs fully) with a total maximum score: 66 points (higher scores, best clinical profile).
Box and Block test (BBT) | Baseline (T0), after 15 rehabilitation sessions (each session is 60 minutes) from 3 to 5 weeks after T0 (T1), 1-month follow-up (T2)
  The Box and Block Test (BBT) measures unilateral gross manual dexterity. The BBT goal is to move, one by one, the maximum number of blocks from one compartment of a box to another of equal size, within 60 seconds. The score is determined by counting the number of blocks carried over the partition from one compartment to the other during the one-minute trial period. Higher scores on the test indicate better gross manual dexterity
EuroQol 5-Dimension 5-level (EQ-5D-5L) Questionnaire | Baseline (T0), after 15 rehabilitation sessions (each session is 60 minutes) from 3 to 5 weeks after T0 (T1), 1-month follow-up (T2)
  EQ-5D-5L is a standardized instrument for use as a measure of health for clinical and economic appraisal. Applicable to a wide range of health conditions and treatments, the EQ-5D health questionnaire provides a simple descriptive profile and a single index value for health status. It measures the 5 dimensions of mobility, self-care, usual activities, pain/discomfort, anxiety/depression. Each dimension is scored on a Likert scale of 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.

SECONDARY OUTCOMES:
Surface Electromyography (EMGs) | Baseline (T0), after 15 rehabilitation sessions (each session is 60 minutes) from 3 to 5 weeks after T0 (T1), 1-month follow-up (T2)
  Surface Electromyography (EMGs) is a non-invasive tool able to assess muscular electrical activity during the execution of active movements using electrodes applied on the skin surface. Muscular contraction amplitude will be recorded from 24 sensors placed on upper limbs (12 sensors/limb), during the execution of motor acts. Then, the difference between patient's and observed model's temporal dynamic of muscular contraction will be chosen as EMG outcome.
Body Kinematics | Baseline (T0), after 15 rehabilitation sessions (each session is 60 minutes) from 3 to 5 weeks after T0 (T1)
  Kinematics of the upper limb and trunk will be recorded using a 9-camera optoelectronic system during 3D motor acts. The system will measure the 3D coordinates of spherical markers attached to body landmarks to compute trunk, shoulder, elbow and wrist angles.
  Data processing will provide measures of deviations from physiological movement.
Treatment Safety | After 15 rehabilitation sessions (each session is 60 minutes) from 3 to 5 weeks after baseline (T1)
  Data related to the safety of the device will be collected:
  1. Number of adverse events
  2. Number of drop-out related to patient intolerance to the device
Cost-effectiveness ratio | At the end of 15 rehabilitation sessions (each session is 60 minutes) from 3 to 5 weeks after baseline (T1)
  The costs of the two rehabilitation paths (with and without device), related to direct costs (maintenance device, consumables) and indirect costs will be collected (training of therapists on the device, costs related to the patient using the device). Procedures to be performed in a single treatment session will also be evaluated, in terms of time needed for preparation and dressing, and of trained personnel required during a session. An estimate of the working cycles that the device can perform in a year will also be considered.

OTHER OUTCOMES:
Age data | Baseline (T0)
  Age of participants will be collected
Gender data | Baseline (T0)
  Gender of participants will be collected
Scholarity data | Baseline (T0)
  Scholarity of participants will be collected

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Ferrarin, PhD, Eng, Principal Investigator — IRCCS Fondazione Don Carlo Gnocchi ONLUS
Locations (3):
- Italy (3):
  - Ospedale Policlinico San Martino, Genova
  - Fondazione Don Carlo Gnocchi Onlus, La Spezia
  - IRCCS Fondazione Don Carlo Gnocchi Onlus, Milan

IPD SHARING:
Plan to Share IPD: Yes
Shared data will comprise only IPD used in results publication. Data will be available upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available after publication with no end date
Access Criteria: Request should be addressed to the principal investigator or the corresponding author of the publication.

REFERENCES:
- [Background] Villepinte C, Verma A, Dimeglio C, De Boissezon X, Gasq D. Responsiveness of kinematic and clinical measures of upper-limb motor function after stroke: A systematic review and meta-analysis. Ann Phys Rehabil Med. 2021 Mar;64(2):101366. doi: 10.1016/j.rehab.2020.02.005. Epub 2020 Mar 7. PMID 32156646
- [Background] de los Reyes-Guzman A, Dimbwadyo-Terrer I, Trincado-Alonso F, Monasterio-Huelin F, Torricelli D, Gil-Agudo A. Quantitative assessment based on kinematic measures of functional impairments during upper extremity movements: A review. Clin Biomech (Bristol). 2014 Aug;29(7):719-27. doi: 10.1016/j.clinbiomech.2014.06.013. Epub 2014 Jun 26. PMID 25017296
- [Background] Roh J, Rymer WZ, Perreault EJ, Yoo SB, Beer RF. Alterations in upper limb muscle synergy structure in chronic stroke survivors. J Neurophysiol. 2013 Feb;109(3):768-81. doi: 10.1152/jn.00670.2012. Epub 2012 Nov 14. PMID 23155178
- [Background] Tropea P, Monaco V, Coscia M, Posteraro F, Micera S. Effects of early and intensive neuro-rehabilitative treatment on muscle synergies in acute post-stroke patients: a pilot study. J Neuroeng Rehabil. 2013 Oct 5;10:103. doi: 10.1186/1743-0003-10-103. PMID 24093623
- [Background] Yang N, An Q, Kogami H, Yamakawa H, Tamura Y, Takahashi K, Kinomoto M, Yamasaki H, Itkonen M, Shibata-Alnajjar F, Shimoda S, Hattori N, Fujii T, Otomune H, Miyai I, Yamashita A, Asama H. Temporal Features of Muscle Synergies in Sit-to-Stand Motion Reflect the Motor Impairment of Post-Stroke Patients. IEEE Trans Neural Syst Rehabil Eng. 2019 Oct;27(10):2118-2127. doi: 10.1109/TNSRE.2019.2939193. Epub 2019 Sep 4. PMID 31494552
- [Background] Overduin SA, d'Avella A, Roh J, Carmena JM, Bizzi E. Representation of Muscle Synergies in the Primate Brain. J Neurosci. 2015 Sep 16;35(37):12615-24. doi: 10.1523/JNEUROSCI.4302-14.2015. PMID 26377453
- [Background] Golicki D, Niewada M, Buczek J, Karlinska A, Kobayashi A, Janssen MF, Pickard AS. Validity of EQ-5D-5L in stroke. Qual Life Res. 2015 Apr;24(4):845-50. doi: 10.1007/s11136-014-0834-1. Epub 2014 Oct 28. PMID 25347978
- [Background] Dorman PJ, Waddell F, Slattery J, Dennis M, Sandercock P. Is the EuroQol a valid measure of health-related quality of life after stroke? Stroke. 1997 Oct;28(10):1876-82. doi: 10.1161/01.str.28.10.1876. PMID 9341688
- [Background] Page SJ, Fulk GD, Boyne P. Clinically important differences for the upper-extremity Fugl-Meyer Scale in people with minimal to moderate impairment due to chronic stroke. Phys Ther. 2012 Jun;92(6):791-8. doi: 10.2522/ptj.20110009. Epub 2012 Jan 26. PMID 22282773
- [Background] Crow JL, Kwakkel G, Bussmann JB, Goos JA, Harmeling-van der Wel BC; Early Prediction of Functional Outcome After Stroke (EPOS) Investigators. Are the hierarchical properties of the Fugl-Meyer assessment scale the same in acute stroke and chronic stroke? Phys Ther. 2014 Jul;94(7):977-86. doi: 10.2522/ptj.20130170. Epub 2014 Mar 27. PMID 24677254
- [Background] Alt Murphy M, Resteghini C, Feys P, Lamers I. An overview of systematic reviews on upper extremity outcome measures after stroke. BMC Neurol. 2015 Mar 11;15:29. doi: 10.1186/s12883-015-0292-6. PMID 25880033
- [Background] van der Lee JH, Beckerman H, Lankhorst GJ, Bouter LM. The responsiveness of the Action Research Arm test and the Fugl-Meyer Assessment scale in chronic stroke patients. J Rehabil Med. 2001 Mar;33(3):110-3. doi: 10.1080/165019701750165916. PMID 11482350
- [Background] Van der Lee JH, De Groot V, Beckerman H, Wagenaar RC, Lankhorst GJ, Bouter LM. The intra- and interrater reliability of the action research arm test: a practical test of upper extremity function in patients with stroke. Arch Phys Med Rehabil. 2001 Jan;82(1):14-9. doi: 10.1053/apmr.2001.18668. PMID 11239280
- [Background] Burton Q, Lejeune T, Dehem S, Lebrun N, Ajana K, Edwards MG, Everard G. Performing a shortened version of the Action Research Arm Test in immersive virtual reality to assess post-stroke upper limb activity. J Neuroeng Rehabil. 2022 Dec 3;19(1):133. doi: 10.1186/s12984-022-01114-3. PMID 36463219
- [Background] Carpinella I, Mazzoleni P, Rabuffetti M, Thorsen R, Ferrarin M. Experimental protocol for the kinematic analysis of the hand: definition and repeatability. Gait Posture. 2006 Jun;23(4):445-54. doi: 10.1016/j.gaitpost.2005.05.001. Epub 2005 Jun 22. PMID 15978812
- [Background] Feng YS, Kohlmann T, Janssen MF, Buchholz I. Psychometric properties of the EQ-5D-5L: a systematic review of the literature. Qual Life Res. 2021 Mar;30(3):647-673. doi: 10.1007/s11136-020-02688-y. Epub 2020 Dec 7. PMID 33284428
- [Background] Chen HM, Chen CC, Hsueh IP, Huang SL, Hsieh CL. Test-retest reproducibility and smallest real difference of 5 hand function tests in patients with stroke. Neurorehabil Neural Repair. 2009 Jun;23(5):435-40. doi: 10.1177/1545968308331146. Epub 2009 Mar 4. PMID 19261767
- [Background] Fugl-Meyer AR, Jaasko L, Leyman I, Olsson S, Steglind S. The post-stroke hemiplegic patient. 1. a method for evaluation of physical performance. Scand J Rehabil Med. 1975;7(1):13-31. PMID 1135616
- [Background] van der Lee JH, Roorda LD, Beckerman H, Lankhorst GJ, Bouter LM. Improving the Action Research Arm test: a unidimensional hierarchical scale. Clin Rehabil. 2002 Sep;16(6):646-53. doi: 10.1191/0269215502cr534oa. PMID 12392340
- [Background] Li L, Scott CA, Rothwell PM. Association of Younger vs Older Ages With Changes in Incidence of Stroke and Other Vascular Events, 2002-2018. JAMA. 2022 Aug 9;328(6):563-574. doi: 10.1001/jama.2022.12759. PMID 35943470
- [Background] Wafa HA, Wolfe CDA, Emmett E, Roth GA, Johnson CO, Wang Y. Burden of Stroke in Europe: Thirty-Year Projections of Incidence, Prevalence, Deaths, and Disability-Adjusted Life Years. Stroke. 2020 Aug;51(8):2418-2427. doi: 10.1161/STROKEAHA.120.029606. Epub 2020 Jul 10. PMID 32646325
- [Background] Winstein CJ, Stein J, Arena R, Bates B, Cherney LR, Cramer SC, Deruyter F, Eng JJ, Fisher B, Harvey RL, Lang CE, MacKay-Lyons M, Ottenbacher KJ, Pugh S, Reeves MJ, Richards LG, Stiers W, Zorowitz RD; American Heart Association Stroke Council, Council on Cardiovascular and Stroke Nursing, Council on Clinical Cardiology, and Council on Quality of Care and Outcomes Research. Guidelines for Adult Stroke Rehabilitation and Recovery: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2016 Jun;47(6):e98-e169. doi: 10.1161/STR.0000000000000098. Epub 2016 May 4. PMID 27145936
- [Background] Thorsen R, Cortesi M, Jonsdottir J, Carpinella I, Morelli D, Casiraghi A, Puglia M, Diverio M, Ferrarin M. Myoelectrically driven functional electrical stimulation may increase motor recovery of upper limb in poststroke subjects: a randomized controlled pilot study. J Rehabil Res Dev. 2013;50(6):785-94. doi: 10.1682/JRRD.2012.07.0123. PMID 24203541
- [Background] Whitehead AL, Julious SA, Cooper CL, Campbell MJ. Estimating the sample size for a pilot randomised trial to minimise the overall trial sample size for the external pilot and main trial for a continuous outcome variable. Stat Methods Med Res. 2016 Jun;25(3):1057-73. doi: 10.1177/0962280215588241. Epub 2015 Jun 19. PMID 26092476
- [Background] Crepaldi M, Thorsen R, Jonsdottir J, Scarpetta S, De Michieli L, Salvo MD, Zini G, Laffranchi M, Ferrarin M. FITFES: A Wearable Myoelectrically Controlled Functional Electrical Stimulator Designed Using a User-Centered Approach. IEEE Trans Neural Syst Rehabil Eng. 2021;29:2142-2152. doi: 10.1109/TNSRE.2021.3120293. Epub 2021 Oct 28. PMID 34648454
- [Background] Jonsdottir J, Thorsen R, Aprile I, Galeri S, Spannocchi G, Beghi E, Bianchi E, Montesano A, Ferrarin M. Arm rehabilitation in post stroke subjects: A randomized controlled trial on the efficacy of myoelectrically driven FES applied in a task-oriented approach. PLoS One. 2017 Dec 4;12(12):e0188642. doi: 10.1371/journal.pone.0188642. eCollection 2017. PMID 29200424
- [Background] Perini G, Bertoni R, Thorsen R, Carpinella I, Lencioni T, Ferrarin M, Jonsdottir J. Sequentially applied myoelectrically controlled FES in a task-oriented approach and robotic therapy for the recovery of upper limb in post-stroke patients: A randomized controlled pilot study. Technol Health Care. 2021;29(3):419-429. doi: 10.3233/THC-202371. PMID 33386831
- [Background] Eraifej J, Clark W, France B, Desando S, Moore D. Effectiveness of upper limb functional electrical stimulation after stroke for the improvement of activities of daily living and motor function: a systematic review and meta-analysis. Syst Rev. 2017 Feb 28;6(1):40. doi: 10.1186/s13643-017-0435-5. PMID 28245858
- [Background] Mehrholz J, Pohl M, Platz T, Kugler J, Elsner B. Electromechanical and robot-assisted arm training for improving activities of daily living, arm function, and arm muscle strength after stroke. Cochrane Database Syst Rev. 2015 Nov 7;2015(11):CD006876. doi: 10.1002/14651858.CD006876.pub4. PMID 26559225
- [Background] Bernhardt J, Hayward KS, Kwakkel G, Ward NS, Wolf SL, Borschmann K, Krakauer JW, Boyd LA, Carmichael ST, Corbett D, Cramer SC. Agreed definitions and a shared vision for new standards in stroke recovery research: The Stroke Recovery and Rehabilitation Roundtable taskforce. Int J Stroke. 2017 Jul;12(5):444-450. doi: 10.1177/1747493017711816. PMID 28697708
- [Background] Raghavan P. Upper Limb Motor Impairment After Stroke. Phys Med Rehabil Clin N Am. 2015 Nov;26(4):599-610. doi: 10.1016/j.pmr.2015.06.008. Epub 2015 Aug 25. PMID 26522900